CLINICAL TRIAL: NCT05209516
Title: Study of Motor Inhibition in Parkinson's Disease and Focal Hand Dystonia (PART 1: Two Parkinson's Disease Projects)
Brief Title: Study of Motor Inhibition in Parkinson's Disease and Focal Hand Dystonia
Acronym: PD-INHIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/27AVR/194
Record Dates: First submitted 2019-07-23; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Surveys and Questionnaires; Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: Three groups of participants: 2 Parkinson patients groups and 1 control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parkinson's disease (PD) patients Group 1 (Experimental): PD patients treated by Dopamine replacement therapy, recruited through Movement Disorders consultations at the Saint-Luc University Hospital, mainly of Prof. Jeanjean, Prof. Ivanoiu, Dr. Wilhelm
  Interventions: Behavioral: Behavioral data; Diagnostic Test: Single-pulse transcranial magnetic stimulation (TMS); Other: Questionnaires; Other: MDS (Movement Disorder Society) UPDRS (Unified Parkinson's Disease Rating Scale) Part 3 (Motor Part)
- Parkinson's disease (PD) patients Group 2 (Experimental): PD patients treated by Deep Brain Stimulation, recruited through Movement Disorders consultations at the Saint-Luc University Hospital, mainly of Prof. Jeanjean, Prof. Ivanoiu, Dr. Wilhelm
  Interventions: Behavioral: Behavioral data; Diagnostic Test: Single-pulse transcranial magnetic stimulation (TMS); Other: Questionnaires; Other: MDS (Movement Disorder Society) UPDRS (Unified Parkinson's Disease Rating Scale) Part 3 (Motor Part)
- Healthy individuals (Active Comparator): Healthy participants, aged between 18 and 85, will be recruited as control subjects by means of ads posting.
  Interventions: Behavioral: Behavioral data; Diagnostic Test: Single-pulse transcranial magnetic stimulation (TMS); Other: Questionnaires

INTERVENTIONS:
Behavioral: Behavioral data — Participants will be seated comfortably in front of a cathode ray tube screen, at a distance of 50-70 cm. The refresh rate of the monitor will be kept above 75 Hz to avoid visual fatigue. Participants will be asked to perform an instructed-delay choice reaction-time task in which they will have to choose between a left and right finger response. In this task, we measure the reaction-times and movement times.
Diagnostic Test: Single-pulse transcranial magnetic stimulation (TMS) — While being comfortably seated in a chair and performing the pre-mentioned task, the participants will undergo single-pulse TMS over both primary motor cortices (M1). In order to guarantee the position of the stimulation coils throughout the testing, participants are asked to wear an EEG cap which will be used to mark various scalp locations. Bipolar surface electrodes, linked to an electromyography (EMG) system, will be placed over one or more muscles of each hand in order to measure the amplitude of motor evoked potentials at various stages of the task. Prior to the placement of each adhesive surface electrode, the skin will be gently swabbed with an alcohol solution.
Other: Questionnaires — Montreal Cognitive Assessment (MoCA), Beck Depression Inventory (BDI) II, Scale on impulsive behaviour (UPPS).
Other: MDS (Movement Disorder Society) UPDRS (Unified Parkinson's Disease Rating Scale) Part 3 (Motor Part) — Specific Parkinson Questionnaire on Clinical motor status
  Arms: Parkinson's disease (PD) patients Group 1; Parkinson's disease (PD) patients Group 2

SUMMARY:
The current research protocol aims at studying preparatory inhibition in two populations of patients suffering from movement disorders. First, in PART 1, we will work with Parkinson's disease (PD) patients to investigate the contribution of the basal ganglia in preparatory inhibition (Project 1 [P1] and Project 2 [P2]). Then, in PART 2, we will consider patients with focal hand dystonia (FHD), to test the hypothesis that altered muscle selectivity in this pathological condition is, at least in part, due to a lack of preparatory inhibition.

DETAILED DESCRIPTION:
Any movement requires some planning, relying substantially on neural cells in the frontal cortex connected with spinal circuits, which themselves help regulating muscle activity. These corticospinal projections provide a critical route through which the brain controls motor behaviour. Interestingly, the excitability of the corticospinal pathway can be investigated non-invasively in humans by applying single-pulse transcranial magnetic stimulation (TMS) over the primary motor cortex (M1), eliciting motor-evoked potentials (MEPs) in targeted contralateral muscles. MEPs are useful indicators of motor excitability, as their amplitude provides a muscle-specific assay of the net impact of facilitatory and inhibitory inputs at the time of the stimulation. Critically, TMS studies have revealed that the corticospinal pathway shows profound inhibitory changes during action preparation, consistent with the contribution of inhibitory processes to movement control.

This effect, referred to as preparatory inhibition, has been evidenced in reaction time (RT) tasks, regardless of whether the subjects have to select a response within a set of predefined options (choice RT task) or have to specify the same response on every trial, in the absence of choice (simple RT task). In these tasks, as expected, the amplitude of MEPs elicited in the selected effector rises during the pre-movement period. However, before activity begins to ramp up, there is an initial decrease in the amplitude of MEPs, indicating the suppression of the corticospinal pathway associated with the selected movement. A reduction in MEP amplitude is also observed in non-selected and irrelevant effectors, and here, the amplitude further drops over the course of action preparation. Preparatory inhibition is not only present preceding movement onset; it is also manifest before the go signal in instructed-delay RT tasks, when a cue provides advance information about the forthcoming response, but the subject must then wait until the go signal is presented to release his response. At that time, suppression is evident for MEPs elicited in finger effectors, including those that are selected, non-selected or task-irrelevant; leg muscle MEPs can also show some suppression during preparation of finger responses but to a much weaker extent , indicating that preparatory inhibition of the motor system is broad, but with some degree of restriction; it is most prominent for motor representations that are from the same body segment as the selected effector and attenuated in other limb representations.

Several hypotheses have been advanced to explain the broad suppression of corticospinal excitability observed during action preparation, with some related to impulse control and others to neural gain modulation. Yet, the functional role of preparatory inhibition remains intensively debated. Further, there is very little knowledge about the brain regions involved in generating this suppression in the corticospinal pathway.

The current research protocol aims at studying preparatory inhibition in two populations of patients suffering from movement disorders. First, we will work with Parkinson's disease (PD) patients to investigate the contribution of the basal ganglia in preparatory inhibition (Project 1 [P1] and Project 2 [P2], see below). Then, we will consider patients with focal hand dystonia (FHD), to test the hypothesis that altered muscle selectivity in this pathological condition is, at least in part, due to a lack of preparatory inhibition (Project 3 [P3], described below).

Beyond its fundamental goals, the present proposal may also provide scientific knowledge to guide intervention strategies that improve motor function in PD and FHD patients. This issue is of great relevance given the increasing life expectancy in our society and the increasing incidence of PD (in particular) that goes with it. The present proposal may also help develop intervention strategies in other pathologies associated with inhibitory deficits, including impulsive decision-making (e.g. PD; drug addiction). This issue is of great importance given the prevalence of such pathologies in our contemporary society.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD (according to the United Kingdom PD Society Brain Bank Clinical Diagnostic Criteria) (for PD participants)
* Good response to levodopa (improvement on the UPDRS-III scale) (for PD participants)
* Hoehn and Yahr stage: < or = 3 (for PD participants)
* Absence of severe tremor (for PD participants)
* Absence of dyskinesia (for PD participants)
* Between 18 and 85 years old (for all participants)
* Normal or corrected-to-normal vision (for all participants)

Exclusion Criteria (for all participants):

* Severe cognitive impairment (Score of <21/30 with the Montreal Cognitive Assessment (MoCA))
* MRI-incompatible metal device in the body
* History of major psychiatric or neurological disorder (other than PD for the patient group)
* Personal or family history of epilepsy
* History of substance use disorder (except nicotine)
* Untreated or unstable medical conditions that could interfere with cognitive functioning
* Undergoing any drug treatment that can significantly alter task performance or neural activity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-04-23 (Estimated); Study Completion 2023-04-23 (Estimated)

PRIMARY OUTCOMES:
TMS measures of preparatory Inhibition | Every participant comes to the laboratory on two consecutive days. All data is acquired on those two days and there are no follow-up measurements. Data acquisition is expected to take up to 6 months per arm.
  TMS is applied while participants are performing the task, either at rest (baseline) or when they are preparing their response (delay).
  Preparatory Inhibition is assessed by expressing MEP amplitudes obtained at TMS-delay relatively to those obtained at TMS-baseline.
  In the present study, Preparatory Inhibition is assessed on two consecutive days in PD patients (ON and OFF dopamine replacement therapy in P1; ON and OFF DBS in P2; randomized order) and healthy control subjects.
Reaction times and movement times during the task | Every participant comes to the laboratory on two consecutive days. All data is acquired on those two days and there are no follow-up measurements. Data acquisition is expected to take up to 6 months per arm.
  The choice RT task allows to measure the reaction and movement times (in ms) for each index finger (left and right), in both PD patients and control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian IVANOIU, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Julie DUQUE, PhD, Study Director — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No